CLINICAL TRIAL: NCT05984758
Title: A Randomised Feasibility Study of Imaging Based Uveitis Screening for Children With Juvenile Idiopathic Arthritis
Brief Title: Imaging Based Uveitis Screening for Children With Juvenile Idiopathic Arthritis
Acronym: UVESCREEN1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21PL04; IRAS (Other: 332422)
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Uveitis, Anterior; Juvenile Idiopathic Arthritis
Keywords: Screening; Surveillance; Imaging; Optical coherence tomography
MeSH Terms: conditions — Uveitis, Anterior; Arthritis, Juvenile | interventions — Slit Lamp Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Active Comparator): Routine examination for uveitis with assessment of visual function followed by slit lamp examination
  Interventions: Diagnostic Test: Slit lamp examination
- ASOCT imaging (Experimental): Assessment of visual function followed by image acquisition with the Optovue RTVue OCT and the Heidelberg Spectralis OCT2 machines
  Interventions: Diagnostic Test: AS-OCT imaging

INTERVENTIONS:
Diagnostic Test: AS-OCT imaging — Image acquisition with the Optovue RTVue OCT and the Heidelberg Spectralis OCT2 machines
  Arms: ASOCT imaging
Diagnostic Test: Slit lamp examination — SLE of anterior chamber
  Arms: Standard care

SUMMARY:
This study seeks to describe, for children undergoing uveitis surveillance following a new diagnosis of juvenile idiopathic arthritis, the feasibility metrics of undertaking a randomised comparative study of routine slit lamp examination (SLE) versus imaging based (anterior segment optical coherence tomography, OCT) surveillance in order to inform the development of a larger multi-centre trial.

DETAILED DESCRIPTION:
This study will compare imaging-based surveillance to routine clinical surveillance for uveitis in children with juvenile idiopathic arthritis (JIA) in order to support the design of a future study.

Childhood uveitis is a rare inflammatory eye disease. Half of all children with uveitis also have a joint disorder: juvenile idiopathic arthritis (or JIA). Children with JIA must travel to a specialist centre every three months to have eye examinations in an attempt to pick uveitis up early enough to prevent visual loss.

Optical coherence tomography (OCT) is a non-contact non-irradiating imaging modality. The investigators have recently demonstrated that novel application of OCT for uveitis detection in children is feasible, acceptable to families, repeatable, sensitive, and specific. The investigators have also found that families welcome the objectivity of imaging-based diagnosis. Standardised operating protocols for image acquisition and analysis have been developed across three imaging platforms (Optovue, Casia and Heidelberg OCT machines).

The investigators will be undertaking a feasibility study which compares routine clinical examination based uveitis surveillance to imaging based surveillance in order to provide the necessary information to address this issue in a larger scale clinical trial of clinical and cost-effectiveness, and explore issues around the impact of objective disease metrics on family perceptions of disease and treatment, as well as the perceptions of children, families and clinical staff on the use of automated diagnostic tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed (within preceding 12 months) with JIA who are eligible for uveitis surveillance
* Aged 2-12 years

Exclusion Criteria:

* A previous / existing diagnosis of uveitis
* Any co-existing ocular or neurological abnormality which impacts on current corrected visual function, or could impact on future corrected visual function
* Developmental/learning difficulties that preclude concordance with examination / informed assent

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who meet the eligibility criteria | 18Months
  Feasibility data for larger scale study
Number of eligible patients recruited | 18Months
  Feasibility data for larger scale study
Proportion of patients that withdraw due to loss of consent or are lost to follow-up | 18Months
  Feasibility data for larger scale study

SECONDARY OUTCOMES:
Success | 12Months
  Success rates (ie agreement with routine clinical examination, set at 100% for routine examination arm, and analysed at 6 months and 12 months milestones for OCT arm)
Pediatric quality of life inventory (PedsQL) child self-report | 12Months
  Health related quality of life, through child self-report, items linearly score on 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life)
Visual analogue scoring (VAS) of examination procedures | 12Months
  Scale running from 0 - 100, with higher score meaning better experience as reported by child

OTHER OUTCOMES:
New diagnoses | 12months
  Number of new diagnoses of uveitis / Number of new diagnosis of other visual/ocular problems

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD shared only after dissemination of study findings and only on reasonable request

REFERENCES:
- [Derived] Dave S, Rahi JS, Petrushkin H, Testi I, Patel DE, Solebo AL. UVESCREEN1: A randomised feasibility study of imaging-based uveitis screening for children with juvenile idiopathic arthritis- Study Protocol. PLoS One. 2025 Feb 12;20(2):e0316410. doi: 10.1371/journal.pone.0316410. eCollection 2025. PMID 39937818